CLINICAL TRIAL: NCT05006404
Title: Autus Size-Adjustable Valve for Surgical Pulmonary Valve Replacement Pivotal Study
Brief Title: Autus Valve Pivotal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Autus Valve Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUT-CP-001
Record Dates: First submitted 2021-07-23; First posted 2021-08-16 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Autus Valve Arm (Experimental): Pulmonary Valve Replacement Surgery with the Autus Valve
  Interventions: Device: Pulmonary Valve Replacement Surgery

INTERVENTIONS:
Device: Pulmonary Valve Replacement Surgery — Pulmonary valve replacement surgery with the Autus Valve

SUMMARY:
Prospective, single-arm, multi-center study to evaluate safety and effectiveness of the Autus Size-Adjustable Valve in pediatric patients aged 18 months to 16 years requiring surgical pulmonary valve replacement. The Autus Valve may be expanded pre-implant to match the subject's body size. Subjects will be evaluated prior to the Autus Valve implant procedure, immediately post-implant, at hospital discharge, 30 days, 6 months, and annually through 10 years.

The Autus Valve may be expanded post-implant via transcatheter balloon dilation to accommodate growth of the subject. In subjects who undergo a post-implant valve expansion, follow-up will continue for a minimum of 1 year after the post-implant valve expansion procedure.

ELIGIBILITY:
Inclusion Criteria:

Candidates must meet all of the following inclusion criteria to be considered for enrollment in this study.

1. Age 18 months to 16 years.
2. Male or female.
3. Subject has a native or repaired right ventricular outflow tract.
4. Subject has been recommended for surgical pulmonary valve replacement by treating clinical team (cardiologist and cardiac surgeon).
5. Subject has at least one of the following echocardiographic findings:

   1. Severe pulmonary stenosis (defined as RV to PA peak instantaneous gradient ≥60 mmHg);
   2. Moderate or greater pulmonary regurgitation;
   3. Moderate or greater pulmonary stenosis plus moderate or greater pulmonary regurgitation.
6. Subject's body size is suitable for implantation of a study device ranging from 12.7 to 22 mm (internal diameter).
7. Subject and parent/legal representative, where appropriate, are willing to provide informed written consent.
8. Subject and parent/legal representative, where appropriate, and treating physician agree that the subject will return for, and comply with, all required study assessments and follow-up visits.

Exclusion Criteria:

Candidates will be excluded from the study if any of the following conditions are met:

1. Subject requires valve replacement in a non-pulmonary position.
2. Subject has a prosthetic valve at other valve position or will need a prosthetic valve at other valve position (i.e., anticipate additional valve replacements needed within 3 years).
3. Subject has pulmonary arterial hypertension (defined as mean PA pressure ≥25 mmHg).
4. Subject has pulmonary atresia and major aortopulmonary collaterals.
5. Subject has significant peripheral pulmonary artery stenosis.
6. Subject has an active infection requiring current systemic antibiotic therapy (if temporary illness, subject may be a candidate 4 weeks after discontinuation of antibiotics).
7. Subject has active endocarditis or a history of infective endocarditis.
8. Subject has renal insufficiency as determined by a serum creatinine (S-Cr) level ≥2.5 mg/dL within 60 days prior to the Screening Visit, or has end-stage renal disease.
9. Subject has leukopenia (defined as a white blood cell (WBC) count <3.5 x 103/µL)
10. Subject has acute or chronic anemia (defined as hemoglobin (Hgb) <10.0 g/dl or 6 mmol/L).
11. Subject has thrombocytopenia (defined as platelet count <50 x 103/µL.
12. Subject has a known hypersensitivity to anticoagulants and antiplatelet drugs.
13. Subject has a known autoimmune disease or receives immunosuppressant and/or immunostimulant drugs that the Investigator or Eligibility Screening Committee (ESC) believes may negatively affect study outcomes.
14. Subject needs emergency cardiac or vascular surgery or intervention.
15. Positive pregnancy test prior to valve implant procedure in female subjects who have had their first menses.
16. Subject has, in the opinion of the Investigator, a life expectancy of less than 5 years.
17. Subject or parent/legal representative refuses blood transfusions.
18. Subject has medical, social or psychosocial factors that, in the opinion of the Investigator or ESC, could impact safety or compliance with study procedures.
19. Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening.

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2036-02-05 (Estimated)

PRIMARY OUTCOMES:
Valve Implantation Primary Safety Endpoint | 30 Days post-valve implantation
  Composite Endpoint: Freedom from a device-related complication through 30 days post-valve implantation as adjudicated by an independent Clinical Events Committee (CEC), including:
  * Death;
  * Valve thrombosis requiring intervention;
  * Symptomatic thromboembolism.
Valve Implantation Primary Effectiveness Endpoint | 6 Months post-valve implantation
  Acceptable hemodynamic performance at 6 months post-valve implantation, as assessed by the Echocardiography Core Laboratory or Clinical Events Committee, defined as:
  * A mean RVOT gradient less than or equal to 40 mmHg and
  * Less than moderate pulmonary regurgitation by transthoracic echo and
  * No Autus Valve reintervention except for valve expansion to address prosthesis-patient mismatch.

OTHER OUTCOMES:
Other Safety Outcome - Composite | 6 months and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following other safety outcome will be evaluated at 6 months, and annually through 10 years post-valve implantation by an independent Clinical Events Committee. The composite outcome includes device-related:
  * Death;
  * Valve thrombosis requiring intervention;
  * Symptomatic thromboembolism.
Other Safety Outcome - Mortality | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Mortality, including: all cause, cardiac-related, procedure-related and device-related
Other Safety Outcome - Valve Thrombosis | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Valve thrombosis
Other Safety Outcome - Thromboembolism | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Thromboembolism
Other Safety Outcome - Cardiac or Valve Intervention | 30 days, 6 months, and annually through a minimum of 510 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Other cardiac or valve intervention (surgical or transcatheter)
Other Safety Outcome - Major Hemorrhage | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Major hemorrhage
Other Safety Outcome - Endocarditis | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Endocarditis
Other Safety Outcome - Hemolysis | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Hemolysis
Other Safety Outcome - Device Explantation | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be evaluated by an independent Clinical Events Committee at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Device explantation
Other Safety Outcome - Adverse Events (AE) | 30 days, 6 months, and annually through a minimum of 10 years and up to 11 years post-valve implantation
  The following measure will be reported at 30 days, 6 months, and annually through 10 years post-valve implantation. Subjects that undergo valve expansion in year 10 after device implantation will be followed for an additional year.
  • Adverse events
Other Safety Outcome - Valve/Stent Fracture | pre-discharge, 12 months, and annually through a minimum of 5 years and up to 6 years post-valve implantation. Subjects that undergo post-implant valve expansion will be evaluated pre-discharge and at 12 months post-valve expansion.
  An independent Medical Reviewer will review post-implant chest x-rays to assess for valve/stent fracture. Chest x-rays will be performed at the following timepoints: post-valve implantation at hospital discharge, and annually through 5 years post-valve implantation. If a post-implant valve expansion procedure is performed, chest x-rays will be performed at hospital discharge and 12 months post-procedure.
Other Effectiveness Outcome - Valve Implant Acute Procedural Success | Immediately Post-Valve Implant Procedure
  To meet the definition of success, all the parameters listed below must be achieved, as assessed by Sites using direct pressure measurements and/or transesophageal echo (TEE):
  * RV to PA peak systolic pressure gradient <40 mmHg (direct pressure measurement);
  * None or trivial pulmonary regurgitation (assessed via TEE);
  * No paravalvular leak (assessed via TEE).
Other Effectiveness Outcome - Pulmonary Regurgitation Grade | Baseline, 30 days, 6 months, and annually through 10 years post-valve implant and 30 days, 6 months, and 12 months post-valve expansion.
  Pulmonary regurgitation grade categorized as none, trivial, mild, moderate, severe as evaluated by the Echo Core Laboratory.
Other Effectiveness Outcome - Pulmonary Stenosis Grade | Baseline, 30 days, 6 months, and annually through 10 years post-valve implant and 30 days, 6 months, and 12 months post-valve expansion.
  Pulmonary stenosis grade categorized as none/trivial, mild, moderate, severe, as evaluated by the Echo Core Laboratory.
Other Effectiveness Outcome - Right Ventricular Measures | Baseline, 30 days, 6 months, and annually through 5 years post-valve implant and 30 days, 6 months, and 12 months post-valve expansion.
  Right ventricular (RV) measures, including RV dimension and strain will be evaluated by the Echo Core Laboratory.
Other Effectiveness Outcome - Left Ventricular Measures | Baseline, 30 days, 6 months, and annually through 10 years post-valve implant and 30 days, 6 months, and 12 months post-valve expansion.
  Left ventricular (LV) measures, including LV ejection fraction and strain will be evaluated by the Echo Core Laboratory.
Other Effectiveness Outcome - Modified Ross Functional Classification | Baseline, 30 days, 6 months, and annually through 10 years post-valve implant and 30 days, 6 months, and 12 months post-valve expansion.
  Modified Ross Functional Class as assessed by the Site Investigators
Other Effectiveness Outcome - PedsQL - Cardiac Module | Baseline, 6 months and annually through 10 years post-valve implantation. Subjects that undergo post-implant valve expansion will be evaluated pre-valve expansion, and at 6 and 12 months post-valve expansion.
  The Pediatric Qualify of Life Inventory (PedsQL) Cardiac Module will be administered by Site Personnel.
Other Post-Implant Valve Expansion Safety Outcome - Composite | 30 days after each post-implant valve expansion procedure
  Composite Endpoint: Freedom from device-related complication through 30 days post-valve expansion as adjudicated by an independent CEC:
  * Death;
  * Extracorporeal membrane oxygenation (ECMO) support;
  * Unplanned intervention (surgical or transcatheter);
  * Major hemorrhage
Other Post-Implant Valve Expansion Effectiveness Outcome - Acute Procedural Success | Immediately after each post-implant valve expansion procedure
  To meet the definition of success, at least one of the parameters listed below must be achieved after each post-implant valve expansion is performed, assessed during the same catheterization procedure:
  * RV to aortic systolic pressure ratio: ≤0.5.
  * Peak-to-peak RV to PA systolic pressure gradient: ≤15 mmHg;
  * Peak-to-peak RV to PA systolic pressure gradient: ≥50% reduction (pre vs post valve expansion).
Other Post-Implant Valve Expansion Effectiveness Outcome - Hemodynamic Performance | 6 months after each post-implant valve expansion procedure
  Clinically acceptable hemodynamic performance at 6 months post-valve expansion procedure, as assessed by the Echo Core Laboratory via TTE, defined as:
  * Less than moderate pulmonary regurgitation (PR) by Doppler echocardiography;
  * Transvalvular gradient (assessed by CW Doppler) at 6-months is lower than the pre-expansion gradient.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie-Charlotte Hofferberth, MD, Study Director — Autus Valve Technologies, Inc.
Locations (12):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan - Mott Children's Hospital, Ann Arbor, Michigan
  - Columbia University Irving Medical Center/New York Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah - Intermountain Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No